CLINICAL TRIAL: NCT05586945
Title: Association of Anemia With Pneumonia in Children up to Two Years Attending Assiut University Children 's Hospital .
Brief Title: Anemia and Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abd Ellatif Ahmed Mohamed, Association of anemia with pneumonia in children up to two years attending AssiutU university children hospital, Assiut University
Other Study IDs: anemia and pneumonia
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess prevalence of anemia among pneumonic children aged two months up to two years.

DETAILED DESCRIPTION:
Pneumonia is an infection via one or both lungs . bacteria and viruses are the most common causes. pneumonia can be medical emergency especially among high risk group like children less than five years Iron deficiency anemia is one of the major health problem in young children. It may be associated with increased risk of pneumonia (1).

A study conducted by Bhaskaram reported high frequency of anemia 83 % in children with pneumonia (2). Iron functions in the immune system are essential, among which are included: the maintenance of the activity of phagocyte oxidase, an iron excess can be used by bacteria to improve its growth (3). Anemia was found to be independently associated with fatal outcome in pneumonic children (4). The risk of development of pneumonia in children with anemia increases approximately by four times in comparison with children who have no anemic syndrome (5).

Breast-feeding protects against lower respiratory tract infection because of breast milk's unique antiinfective properties (6). Infants who were not being breast fed were 17 times more likely than those being breast fed without formula milk to be admitted to hospital for pneumonia (7). one of the factors that affects severe malnutrition is wrong parenting as parents can play an important role in their children's growth through proper, adequate feeding (8). There's no available studies that examine the association between anemia and pneumonia in our locality.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria: Children aged two months up to two years who attend to Assiut University Hospital with pneumonia in the outpatient pediatric clinic, emergency unit and from inpatient .

Exclusion Criteria:

* . Exclusion criteria: All patients with other comorbidities will be excluded from our study as: severe sepsis & localized infection e.g endocarditis, empyema, autoimmune diseases,renal diseases and congenital anomaly

Ages: 2 Months to 2 Years | Sex: All
Age Groups: Child
Study Population: Children aged 2 month S up to two years
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Determine association between anemia and pneumonia in children aged two months up to two years Secondary (subsidiary): Study other associated factors as nutrition and sociodemographic factors | 6 months duration